CLINICAL TRIAL: NCT01657682
Title: A Phase II Study of Crenolanib in Relapsed/Refractory Acute Myeloid Leukemia Patients With FLT3 Activating Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARO-005
Record Dates: First submitted 2012-07-31; First posted 2012-08-06 (Estimated); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia With FLT3 Activating Mutations That Has Relapsed or Been Refractory After One or More Prior Therapies
Keywords: FLT3; Crenolanib; Acute; Myeloid; AML

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A - No prior FLT3 TKI exposure (Experimental): Will enroll relapsed/refractory AML patients with FLT3 activating mutations who progressed on one or more prior chemotherapy regimens excluding any FLT3 TKI.
  Interventions: Drug: Crenolanib besylate
- Cohort B - Prior therapy with FLT3 TKI (Experimental): Will enroll relapsed/refractory AML patients with FLT3 activating mutations whose leukemia has progressed and have history of prior therapy with one or more FLT3 TKIs.
  Interventions: Drug: Crenolanib besylate

INTERVENTIONS:
Drug: Crenolanib besylate — Crenolanib besylate, 100 mg TID, taken orally at least 30 minutes pre- or post- meal. Patients will complete a daily diary to record the date, time and amount (number of tablets) of crenolanib taken and eating schedule.
  Concurrent hydroxyurea (maximum 5g total daily dose x 14 days) is permitted during the first 28 days of study therapy.

SUMMARY:
This pilot Phase II study is designed to evaluate the efficacy and tolerability of crenolanib in two cohorts of AML patients with FLT3 activation mutations (patients whose leukemia has recurred after prior chemotherapy not including a FLT3 TKI and patients whose leukemia has progressed after prior therapy with a FLT3 TKI).

DETAILED DESCRIPTION:
This is a Phase II open label study of crenolanib besylate. This study will enroll subjects with relapsed acute myeloid leukemia (AML) with FLT3 activating mutations. Two cohorts of patients will be enrolled: those whose AML has recurred after prior chemotherapy without a FLT3 TKI, and those whose AML has progressed after prior therapy with FLT3 TKIs. Subjects will take Crenolanib besylate at 100 mg TID until disease progression, death, or unacceptable toxicities. Concurrent hydroxyurea is permitted during the first 28 days of study therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary AML relapsed or refractory after prior therapy, AML secondary to antecedent chemotherapy or radiation therapy, or AML due to prior myelodysplastic syndrome (MDS)/ myeloproliferative neoplasm (MPN) as defined by WHO criteria with presence of either FLT3 ITD and/or other FLT3 activating mutations
* Patients with secondary AML should have failed no more than two (2) prior regimens
* Patients with antecedent MDS/MPN, defined by WHO criteria, without any prior therapy for AML, regardless of the number of therapies for MDS/ MPN
* Patients with primary AML should have received no more than two (2) prior cytotoxic containing salvage regimens. Reinduction with the same regimen or stem cell transplant will not be considered a separate salvage regimen. Change of drugs will be considered a salvage regimen. Unlimited FLT3 TKI therapy (even in combination with cytotoxics/hypomethylating agents) is allowed for patients enrolled in cohort B
* Patients must have tested positive for FLT3-ITD and /or other FLT3 activating mutations within 30 day screening period
* Males and females age ≥18 years
* ECOG PS 0-2
* Adequate liver function, defined as bilirubin ≤1.5x ULN, ALT ≤3.0x ULN, and AST ≤3.0x ULN
* Adequate renal function, defined as serum creatinine ≤1.5x ULN
* Recovery from non-hematological toxicities of prior therapy (including HSCT) to no more than grade 1 (except alopecia)
* Subjects should have received no anti-leukemic therapy (except hydroxyurea) prior to the first dose of crenolanib as follows: for 14 days for classical cytotoxic agents and for five times the t1/2 (half-life) for FLT3 inhibitors and antineoplastic agents that are neither cytotoxic nor FLT3 inhibitors (e.g. hypomethylating agent or MEK inhibitor)
* Negative pregnancy test for WOCBP
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Absence of a FLT3 activating mutation
* <5% blasts in blood or marrow at screening
* Concurrent chemotherapy, or targeted anti-cancer agents, other than hydroxyurea
* Patient with concurrent severe and/or uncontrolled medical conditions that in the opinion of the investigator may impair the participation in the study or the evaluation of safety and/or efficacy
* HIV infection or active hepatitis B (defined as hepatitis B surface antigen positive) or C (defined as hepatitis C antibody positive)
* Known clinically active central nervous system (CNS) leukemia
* Patients less than 30 days post HSCT
* Subjects who have clinically significant graft versus host disease requiring treatment and /or have >grade 2 persistent non hematological toxicity related to transplant
* Prior crenolanib treatment for a non-leukemic indication
* Major surgical procedures within 14 days of Day 1 administration of crenolanib.
* Unwillingness or inability to comply with protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Galanis A, Ma H, Rajkhowa T, Ramachandran A, Small D, Cortes J, Levis M. Crenolanib is a potent inhibitor of FLT3 with activity against resistance-conferring point mutants. Blood. 2014 Jan 2;123(1):94-100. doi: 10.1182/blood-2013-10-529313. Epub 2013 Nov 13. PMID 24227820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 participants who met all inclusion criteria and none of the exclusion criteria were included in the study and were enrolled at 1 center in the United States.
Groups:
- Cohort A - No Prior FLT3 TKI Exposure: Participants who had relapsed/refractory AML with FLT3 activating mutations who progressed on one or more prior chemotherapy regimens excluding any FLT3 TKI received 100 mg crenolanib besylate tablets administered orally three times a day.
- Cohort B - Prior Therapy With FLT3 TKI: Participants who had relapsed/refractory AML with FLT3 activating mutations whose leukemia progressed and have history of prior therapy with one or more FLT3 TKIs received 100 mg crenolanib besylate tablets administered orally three times a day.
- Cohort C - Antecedent Hematological Disorder: Participants who had relapsed/refractory AML with FLT3 activating mutations whose leukemia progressed and have history of antecedent hematological disorder received 100 mg crenolanib besylate tablets administered orally three times a day.
Period: Overall Study
Arm/Group | Cohort A - No Prior FLT3 TKI Exposure | Cohort B - Prior Therapy With FLT3 TKI | Cohort C - Antecedent Hematological Disorder
Started | 13 | 30 | 13
Completed | 12 | 28 | 12
Not Completed | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - No Prior FLT3 TKI Exposure | Cohort B - Prior Therapy With FLT3 TKI | Cohort C - Antecedent Hematological Disorder | Total
Number analyzed (Participants) | 13 | 30 | 13 | 56
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 44 years | 2 | 7 | 2 | 11
  Between 45 and 60 years | 4 | 8 | 3 | 15
  >60 years | 7 | 15 | 8 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 7 | 30
  Male | 5 | 15 | 6 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race data was not available for one patient in cohort B.
  Participants
    Race: number analyzed (Participants) | 13 | 29 | 13 | 55
    Race: Black or African American | 0 | 2 | 1 | 3
    Race: Asian | 1 | 5 | 1 | 7
    Race: White | 11 | 18 | 11 | 40
    Race: Other | 1 | 4 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 4 | 0 | 5
  Ethnicity: Not Hispanic or Latino | 12 | 25 | 13 | 50
  Ethnicity: Unknown | 0 | 1 | 0 | 1
Baseline FLT3 mutation [Count of Participants; unit: Participants]
  FLT3-ITD only | 8 | 15 | 3 | 26
  FLT3-TKD only | 5 | 2 | 4 | 11
  FLT3-ITD and FLT3-TKD | 0 | 13 | 6 | 19
Baseline ECOG Performance [Count of Participants; unit: Participants]
  0 - Normal activity | 2 | 3 | 1 | 6
  1 - Symptoms but ambulatory | 9 | 21 | 9 | 39
  2 - In bed < 50% of time | 2 | 6 | 3 | 11
Number of Prior Therapies [Median (Full Range); unit: prior therapies] | 2 [1 to 4] | 3 [1 to 6] | 2 [1 to 6] | 3 [1 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Patients Receiving Crenolanib Therapy
Description: To determine the response rate to crenolanib. CR Complete remission (CR) response criteria include a post-baseline bone marrow (BM) biopsy or aspiration % blasts <5%, absolute neutrophil count (ANC) >1×10^9/L and platelet count >100×10^9/L. CRi response included all CR criteria met, except participant did not experience either platelet recovery or ANC recovery. Partial Response (PR) response included a decrease of ≥50% in % blasts in the BM aspirate or biopsy from baseline to a post-baseline result between 5% to 25% in the bone marrow aspirate or biopsy. Blast reduction (BR) response included a decrease of ≥50% in % blasts. Resistant Disease (RD) was defined as the absence of CR, CRi, CRp, PR or MLFS.
Time Frame: From the date of first dose to the end of protocol treatment.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: Participants who had relapsed/refractory AML with FLT3 activating mutations who progressed on one or more prior chemotherapy regimens received 100 mg crenolanib besylate tablets administered orally three times a day.
Arm/Group | All Patients | Cohort A - No Prior FLT3 TKI Exposure | Cohort B - Prior Therapy With FLT3 TKI | Cohort C - Antecedent Hematological Disorder
Number analyzed (Participants) | 56 | 13 | 30 | 13
Participants
  CR/CRi | 8 | 3 | 4 | 1
  PR | 9 | 2 | 5 | 2
  ORR (CR+PR) | 17 | 5 | 9 | 3
  BR | 21 | 5 | 11 | 5
  Clinical Benefit (CR+PR+BR) | 38 | 10 | 20 | 8
  Resistant disease (RD) | 18 | 3 | 10 | 5

2. Secondary Outcome: Duration of Overall Survival
Description: To determine the overall survival of AML patients with activating FLT3 mutations treated with crenolanib
Time Frame: From the date of first dose up to end of treatment, up to 24 months.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A - No Prior FLT3 TKI Exposure | Cohort B - Prior Therapy With FLT3 TKI | Cohort C - Antecedent Hematological Disorder
Number analyzed (Participants) | 13 | 30 | 13
days | 237 [134 to 548] | 100 [76 to 192] | 85 [49 to 329]

3. Secondary Outcome: Study Drug Exposure
Description: To determine the study drug exposure of relapse/refractory AML patients receiving 100 mg crenolanib besylate tablets three times daily.
Time Frame: Defined as the duration from first day to the last dose, up to 24 months, interruptions in study drug administration were not counted.
Measure: Median (Full Range); unit: days
Groups:
- Cohort A - No Prior FLT3 TKI Exposure: Participants who had relapsed/refractory AML with FLT3 activating mutations whose leukemia progressed on one or more prior chemotherapy regimens excluding any FLT3 TKI received 100 mg crenolanib besylate tablets administered orally three times a day.
- Cohort B - Prior Therapy With FLT3 TKI: Participants who had relapsed/refractory AML with FLT3 activating mutations whose leukemia progressed on one or more prior chemotherapy regimens and have history of prior therapy with one or more FLT3 TKI received 100 mg crenolanib besylate tablets administered orally three times a day.
- Cohort C - Antecedent Hematological Disorder: Participants who had relapsed/refractory AML with FLT3 activating mutations whose leukemia progressed on one or more prior chemotherapy regimens and have history of antecedent hematological disorder received 100 mg crenolanib besylate tablets administered orally three times a day.
Arm/Group | Cohort A - No Prior FLT3 TKI Exposure | Cohort B - Prior Therapy With FLT3 TKI | Cohort C - Antecedent Hematological Disorder
Number analyzed (Participants) | 13 | 30 | 13
days | 57 [16 to 139] | 43.5 [5 to 197] | 50 [10 to 138]

ADVERSE EVENTS:
Time Frame: From the date of first dose up to end of treatment, up to 24 months.
Arm/Group | All Patients | Cohort A - No Prior FLT3 TKI Exposure | Cohort B - Prior Therapy With FLT3 TKI | Cohort C - Antecedent Hematological Disorder
All-Cause Mortality (participants affected / at risk) | 53/56 | 12/13 | 29/30 | 12/13
Serious Adverse Events (participants affected / at risk) | 52/56 | 10/13 | 30/30 | 12/13
Other Adverse Events (participants affected / at risk) | 56/56 | 13/13 | 30/30 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=56) | Cohort A - No Prior FLT3 TKI Exposure (N=13) | Cohort B - Prior Therapy With FLT3 TKI (N=30) | Cohort C - Antecedent Hematological Disorder (N=13)
Anemia (Blood and lymphatic system disorders) | 4 | 1 | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 4 | 8 | 3
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 3 | 0 | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 4 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 5 | 0 | 4 | 1
Nausea (Gastrointestinal disorders) | 4 | 0 | 2 | 2
Parotitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 2 | 1
Mouth hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Death (General disorders) | 4 | 1 | 2 | 1
Disease progression (General disorders) | 6 | 1 | 5 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0
Generalized edema (General disorders) | 1 | 0 | 1 | 0
Multi-organ failure (General disorders) | 2 | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Edema peripheral (General disorders) | 1 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 1 | 0
Medical device site joint infection (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 18 | 2 | 9 | 7
Pneumonia fungal (Infections and infestations) | 2 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
BK virus infection (Infections and infestations) | 1 | 0 | 1 | 0
Cytomegalovirus viremia (Infections and infestations) | 1 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Oral infection (Infections and infestations) | 1 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 1 | 0
Stenotrophomonas sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 2 | 0 | 0
Hemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0
Cystitis hemorrhagic (Renal and urinary disorders) | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 4 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Anorectal cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hemorrhage (Vascular disorders) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 4 | 2 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Embolism (Vascular disorders) | 1 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=56) | Cohort A - No Prior FLT3 TKI Exposure (N=13) | Cohort B - Prior Therapy With FLT3 TKI (N=30) | Cohort C - Antecedent Hematological Disorder (N=13)
Anaemia (Blood and lymphatic system disorders) | 11 | 4 | 6 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 4 | 8 | 5
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 4 | 0 | 4 | 0
Splenomegaly (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 2 | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 6 | 0 | 5 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 7 | 1 | 4 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 1 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 1 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 1
Erythema of eyelid (Eye disorders) | 1 | 0 | 1 | 0
Eye discharge (Eye disorders) | 1 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 4 | 2 | 2 | 0
Pupils unequal (Eye disorders) | 1 | 0 | 1 | 0
Vision blurred (Eye disorders) | 2 | 0 | 1 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 1 | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 6 | 1 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 32 | 7 | 15 | 10
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 3 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Asthenia (General disorders) | 4 | 0 | 2 | 2
Chest pain (General disorders) | 5 | 1 | 2 | 2
Chills (General disorders) | 5 | 1 | 3 | 1
Death (General disorders) | 4 | 1 | 2 | 1
Disease progression (General disorders) | 7 | 2 | 5 | 0
Face oedema (General disorders) | 3 | 0 | 3 | 0
Fatigue (General disorders) | 25 | 5 | 13 | 7
Gait disturbance (General disorders) | 1 | 0 | 1 | 0
Generalised oedema (General disorders) | 2 | 1 | 1 | 0
Inflammation (General disorders) | 1 | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 3 | 1 | 2 | 0
Multi-organ failure (General disorders) | 2 | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1 | 0
Nodule (General disorders) | 1 | 1 | 0 | 0
Oedema (General disorders) | 4 | 3 | 0 | 1
Oedema mucosal (General disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 22 | 5 | 11 | 6
Pain (General disorders) | 2 | 0 | 1 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 6 | 2 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 6 | 1 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 4 | 2 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 0 | 6 | 1
Gingival bleeding (Gastrointestinal disorders) | 4 | 2 | 2 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 0 | 2 | 2
Lip dry (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Lip exfoliation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 5 | 1 | 2 | 2
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 44 | 11 | 22 | 11
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Parotitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 1 | 3 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 28 | 7 | 16 | 5
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 1 | 1
Graft versus host disease (Immune system disorders) | 1 | 0 | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0
BK virus infection (Infections and infestations) | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 4 | 1 | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 0 | 1 | 1
Enterococcal infection (Infections and infestations) | 1 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Eye infection (Infections and infestations) | 1 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 2 | 1 | 1 | 0
Localised infection (Infections and infestations) | 1 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1 | 0
Medical device site joint infection (Infections and infestations) | 1 | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 2 | 2 | 0 | 0
Oral infection (Infections and infestations) | 1 | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 21 | 2 | 11 | 8
Pneumonia fungal (Infections and infestations) | 3 | 1 | 2 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 2 | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Septic shock (Infections and infestations) | 2 | 0 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1 | 0 | 0
Stenotrophomonas sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Alanine aminotransferase (Investigations) | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2 | 2 | 0
Amylase increased (Investigations) | 1 | 1 | 0 | 0
Aspartate aminotransferase (Investigations) | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0
Blood bilirubin (Investigations) | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 5 | 2 | 3 | 0
Blood creatinine (Investigations) | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 0 | 2 | 1
Blood phosphorus increased (Investigations) | 1 | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0 | 0
Gamma-glutamyltransferase (Investigations) | 2 | 0 | 2 | 0
Lipase increased (Investigations) | 1 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 1 | 0
Pancreatic enzymes increased (Investigations) | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 4 | 1 | 1 | 2
Transaminases increased (Investigations) | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 2 | 0 | 2 | 0
Weight increased (Investigations) | 5 | 1 | 3 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0
White blood cell count increased (Investigations) | 7 | 2 | 4 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 1 | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 7 | 1 | 6 | 0
Fluid overload (Metabolism and nutrition disorders) | 3 | 0 | 1 | 2
Fluid retention (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 2 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 2 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 3 | 5 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 3 | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 3 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 2
Cerebellar ataxia (Nervous system disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 7 | 1 | 6 | 0
Dysgeusia (Nervous system disorders) | 6 | 2 | 2 | 2
Dystonia (Nervous system disorders) | 1 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 2 | 4 | 2
Lethargy (Nervous system disorders) | 2 | 0 | 2 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 1 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 4 | 4 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0
Claustrophobia (Psychiatric disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 5 | 0 | 4 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 3 | 0 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 2 | 1
Bladder dilatation (Renal and urinary disorders) | 1 | 0 | 1 | 0
Bladder pain (Renal and urinary disorders) | 1 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 6 | 2
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 7 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 8 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 1 | 10 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2 | 2
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 4 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Tracheal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Anorectal cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 4 | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0 | 4 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 2
Hypotension (Vascular disorders) | 6 | 3 | 3 | 2
Paraesthenia (Nervous system disorders) | 2 | 1 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT01657682/Prot_SAP_000.pdf